CLINICAL TRIAL: NCT02135250
Title: Study on Therapeutic Effect of Treating Mental Stress Induced Myocardial Ischemia With Conventional Therapy for Coronary Heart Disease Combined With Traditional Chinese Medicine :Design and Methods
Brief Title: Study on Therapeutic Effect of Treating Mental Stress Induced Myocardial Ischemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meiyan Liu (Other)
Responsible Party: Sponsor-Investigator, Meiyan Liu, physician, Beijing Anzhen Hospital
Organization: Beijing Anzhen Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013022
Record Dates: First submitted 2014-05-06; First posted 2014-05-09 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Theraphy of Chinese Traditional Medicine
Keywords: Traditional Chinese Medicine
MeSH Terms: interventions — xinkeshu

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Experimental): the placebo is not drug
  Interventions: Other: placebo
- Xinkeshu tablet (Experimental): 4 Xinkeshu tablets are given three times per day
  Interventions: Drug: Xinkeshu tablets

INTERVENTIONS:
Drug: Xinkeshu tablets — 4 Xinkeshu tablets are given three times per day
  Arms: Xinkeshu tablet
Other: placebo — the placebo is not drug.
  Arms: placebo

SUMMARY:
This study aims to discuss whether the combined treatment of traditional Chinese medicine (TCM) and western medicine for Mental Stress Induced Myocardial Ischemia (MSIMI) does effect, namely the conventional therapy for Coronary Heart Disease( CHD) combining with TCM - Xinkeshu tablets.

DETAILED DESCRIPTION:
A large number of evidence-based medical researches have proven that bad mood and mental stress are related to poor prognosis. Having recognized that acute emotional stress can induce cardiovascular events, many clinical tests of mental stress have been carried out to observe the correlation between emotional stress and cardiac damage, which ultimately lead to the formalization of the concept of Mental Stress Induced Myocardial Ischemia(MSIMI). In the past 3 decades, it has been evidenced that mental stress is internally related to myocardial ischemia. According to current studies, over 70% patients with stable coronary heart disease have MSIMI and are exposed to three or four times higher risk of cardiovascular events. However, few articles are about the therapeutic effect of MSIMI treatment. This study aims to discuss whether the combined treatment of traditional Chinese medicine (TCM) and western medicine for MSIMI does effect, namely the conventional therapy for CHD combining with TCM - Xinkeshu tablets.

ELIGIBILITY:
Inclusion Criteria:

1. above 18 years old,
2. having coronary stenosis (> 70%) measured by coronary arteriography,
3. with medical history of myocardial infarction or revascularization procedures,
4. or with sufficient proof for having CHD.

Exclusion Criteria:

1. patient age younger than 18,
2. clearly impaired cognitive function,
3. damage of functions of vital organs,
4. suicidal ideation,
5. mental diseases treated with selective serotonin reuptake inhibitor (SSRI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction | up to 8 weeks
  reduction of LVEF by 5% or more
ventricular wall motion | up to 8 weeks
  Echocardiography to assess the ventricular wall motion in one cardiac cycle starting from the systole

CONTACTS AND LOCATIONS:
Overall Officials: Anzhen Beijing, Principal Investigator — Capital Medical University
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Faxon DP, Creager MA, Smith SC Jr, Pasternak RC, Olin JW, Bettmann MA, Criqui MH, Milani RV, Loscalzo J, Kaufman JA, Jones DW, Pearce WH; American Heart Association. Atherosclerotic Vascular Disease Conference: Executive summary: Atherosclerotic Vascular Disease Conference proceeding for healthcare professionals from a special writing group of the American Heart Association. Circulation. 2004 Jun 1;109(21):2595-604. doi: 10.1161/01.CIR.0000128517.52533.DB. No abstract available. PMID 15173041
- [Background] Strike PC, Steptoe A. Systematic review of mental stress-induced myocardial ischaemia. Eur Heart J. 2003 Apr;24(8):690-703. doi: 10.1016/s0195-668x(02)00615-2. No abstract available. PMID 12713764
- [Background] Jiang W, Babyak M, Krantz DS, Waugh RA, Coleman RE, Hanson MM, Frid DJ, McNulty S, Morris JJ, O'Connor CM, Blumenthal JA. Mental stress--induced myocardial ischemia and cardiac events. JAMA. 1996 Jun 5;275(21):1651-6. doi: 10.1001/jama.275.21.1651. PMID 8637138
- [Background] Sheps DS, McMahon RP, Becker L, Carney RM, Freedland KE, Cohen JD, Sheffield D, Goldberg AD, Ketterer MW, Pepine CJ, Raczynski JM, Light K, Krantz DS, Stone PH, Knatterud GL, Kaufmann PG. Mental stress-induced ischemia and all-cause mortality in patients with coronary artery disease: Results from the Psychophysiological Investigations of Myocardial Ischemia study. Circulation. 2002 Apr 16;105(15):1780-4. doi: 10.1161/01.cir.0000014491.90666.06. PMID 11956119
- [Background] Liu Y, Huang Y, Zhao C, Qin X, Zhu Q, Chen S, Qu J. Salvia miltiorrhiza injection on pulmonary heart disease: a systematic review and meta-analysis. Am J Chin Med. 2014;42(6):1315-31. doi: 10.1142/S0192415X14500827. PMID 25395310
- [Background] Zhong LY, Shen ZY, Cai DF. [Effect of three kinds (tonifying kidney, invigorating spleen, promoting blood circulation) recipes on the hypothalamus-pituitary-adrenal-thymus (HPAT) axis and CRF gene expression]. Zhongguo Zhong Xi Yi Jie He Za Zhi. 1997 Jan;17(1):39-41. Chinese. PMID 9812651
- [Background] Gao Y, Zhang K, Zhu F, Wu Z, Chu X, Zhang X, Zhang Y, Zhang J, Chu L. Salvia miltiorrhiza (Danshen) inhibits L-type calcium current and attenuates calcium transient and contractility in rat ventricular myocytes. J Ethnopharmacol. 2014 Dec 2;158 Pt A:397-403. doi: 10.1016/j.jep.2014.10.049. Epub 2014 Oct 31. PMID 25446591
- [Background] Maji AK, Pandit S, Banerji P, Banerjee D. Pueraria tuberosa: a review on its phytochemical and therapeutic potential. Nat Prod Res. 2014;28(23):2111-27. doi: 10.1080/14786419.2014.928291. Epub 2014 Jul 1. PMID 24980468
- [Background] Zhao S, Zheng MX, Chen HE, Wu CY, Wang WT. Effect of panax notoginseng saponins injection on the p38MAPK pathway in lung tissue in a rat model of hypoxic pulmonary hypertension. Chin J Integr Med. 2015 Feb;21(2):147-51. doi: 10.1007/s11655-014-1790-2. Epub 2014 Dec 19. PMID 25523598
- [Background] Huang SS, Deng JS, Lin JG, Lee CY, Huang GJ. Anti-inflammatory effects of trilinolein from Panax notoginseng through the suppression of NF-kappaB and MAPK expression and proinflammatory cytokine expression. Am J Chin Med. 2014;42(6):1485-506. doi: 10.1142/S0192415X14500931. PMID 25482678
- [Background] Ghanbari-Niaki A, Ghanbari-Abarghooi S, Rahbarizadeh F, Zare-Kookandeh N, Gholizadeh M, Roudbari F, Zare-Kookandeh A. Heart ABCA1 and PPAR- alpha Genes Expression Responses in Male rats: Effects of High Intensity Treadmill Running Training and Aqueous Extraction of Black Crataegus-Pentaegyna. Res Cardiovasc Med. 2013 Nov;2(4):153-9. doi: 10.5812/cardiovascmed.13892. Epub 2013 Oct 28. PMID 25478513
- [Background] Coulter SA, Campos K. Identify and treat depression for reduced cardiac risk and improved outcomes. Tex Heart Inst J. 2012;39(2):231-4. PMID 22740739
- [Background] Goldberg AD, Becker LC, Bonsall R, Cohen JD, Ketterer MW, Kaufman PG, Krantz DS, Light KC, McMahon RP, Noreuil T, Pepine CJ, Raczynski J, Stone PH, Strother D, Taylor H, Sheps DS. Ischemic, hemodynamic, and neurohormonal responses to mental and exercise stress. Experience from the Psychophysiological Investigations of Myocardial Ischemia Study (PIMI). Circulation. 1996 Nov 15;94(10):2402-9. doi: 10.1161/01.cir.94.10.2402. PMID 8921780
- [Background] Jain D, Shaker SM, Burg M, Wackers FJ, Soufer R, Zaret BL. Effects of mental stress on left ventricular and peripheral vascular performance in patients with coronary artery disease. J Am Coll Cardiol. 1998 May;31(6):1314-22. doi: 10.1016/s0735-1097(98)00092-8. PMID 9581726
- [Background] Kop WJ, Krantz DS, Howell RH, Ferguson MA, Papademetriou V, Lu D, Popma JJ, Quigley JF, Vernalis M, Gottdiener JS. Effects of mental stress on coronary epicardial vasomotion and flow velocity in coronary artery disease: relationship with hemodynamic stress responses. J Am Coll Cardiol. 2001 Apr;37(5):1359-66. doi: 10.1016/s0735-1097(01)01136-6. PMID 11300447
- [Background] Schoder H, Silverman DH, Campisi R, Sayre JW, Phelps ME, Schelbert HR, Czernin J. Regulation of myocardial blood flow response to mental stress in healthy individuals. Am J Physiol Heart Circ Physiol. 2000 Feb;278(2):H360-6. doi: 10.1152/ajpheart.2000.278.2.H360. PMID 10666065
- [Background] Schoder H, Silverman DH, Campisi R, Karpman H, Phelps ME, Schelbert HR, Czernin J. Effect of mental stress on myocardial blood flow and vasomotion in patients with coronary artery disease. J Nucl Med. 2000 Jan;41(1):11-6. PMID 10647599
- [Background] Boushey CJ, Beresford SA, Omenn GS, Motulsky AG. A quantitative assessment of plasma homocysteine as a risk factor for vascular disease. Probable benefits of increasing folic acid intakes. JAMA. 1995 Oct 4;274(13):1049-57. doi: 10.1001/jama.1995.03530130055028. PMID 7563456
- [Background] Woo KS, Sanderson JE, Sun YY, Chook P, Cheung AS, Chan LT, Metreweli C, Lolin YI, Celermajer DS. Hyperhomocyst(e)inemia is a risk factor for arterial endothelial dysfunction in humans. Circulation. 2000 Mar 28;101(12):E116. doi: 10.1161/01.cir.101.12.e116. No abstract available. PMID 10736298
- [Background] Laaksonen R, Janatuinen T, Vesalainen R, Lehtimaki T, Elovaara I, Jaakkola O, Jokela H, Laakso J, Nuutila P, Punnonen K, Raitakari O, Saikku P, Salminen K, Knuuti J. High oxidized LDL and elevated plasma homocysteine contribute to the early reduction of myocardial flow reserve in healthy adults. Eur J Clin Invest. 2002 Nov;32(11):795-802. doi: 10.1046/j.1365-2362.2002.01051.x. PMID 12423319
- [Background] Morrow DA, Cannon CP, Jesse RL, Newby LK, Ravkilde J, Storrow AB, Wu AH, Christenson RH; National Academy of Clinical Biochemistry. National Academy of Clinical Biochemistry Laboratory Medicine Practice Guidelines: Clinical characteristics and utilization of biochemical markers in acute coronary syndromes. Circulation. 2007 Apr 3;115(13):e356-75. doi: 10.1161/CIRCULATIONAHA.107.182882. Epub 2007 Mar 23. No abstract available. PMID 17384331
- [Background] de Lemos JA, Drazner MH, Omland T, Ayers CR, Khera A, Rohatgi A, Hashim I, Berry JD, Das SR, Morrow DA, McGuire DK. Association of troponin T detected with a highly sensitive assay and cardiac structure and mortality risk in the general population. JAMA. 2010 Dec 8;304(22):2503-12. doi: 10.1001/jama.2010.1768. PMID 21139111
- [Background] Bass A, Patterson JH, Adams KF Jr. Perspective on the clinical application of troponin in heart failure and states of cardiac injury. Heart Fail Rev. 2010 Jul;15(4):305-17. doi: 10.1007/s10741-008-9124-8. Epub 2009 Apr 5. PMID 19347578